CLINICAL TRIAL: NCT07096076
Title: Comparison of The Immediate Effects of Thoracolumbar Fascia Inhibition and Suboccipital Muscle Inhibition on Cervical and Lumbar Joint Range of Motion, Flexibility of Back Extensors and Hamstring Muscles, Functional Exercise Capacity, and Balance In Individuals With Hamstring Shortness
Brief Title: The Immediate Effects Of Thoracolumbar Fascia Inhibition And Suboccipital Muscle Inhibition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Sanem ŞENER, Assistant Professor, Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCTHamstring-shortness
Record Dates: First submitted 2025-03-25; First posted 2025-07-31 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Healthy Individuals With Hamstring Tightness

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator)
  Interventions: Other: hamstring stretching
- Thoracolumbar fascia inhibition group (Experimental)
  Interventions: Other: Thoracolumbar fascia inhibition; Other: hamstring stretching
- Suboccipital inhibition group (Experimental)
  Interventions: Other: Suboccipital inhibition group; Other: hamstring stretching

INTERVENTIONS:
Other: Thoracolumbar fascia inhibition — Soft tissue mobilization: Participants will be asked to lie on their backs without a pillow in a hook-lying position, placing a foam roller under the inferior part of the scapula and clasping their hands behind the cervical region. Then, they will be instructed to lift their hips off the ground and roll the foam roller in a cranial and caudal direction from the inferior scapular region to the sacral area for 30 seconds, performing flexion and extension movements with their knees. This application will be performed in a total of 4 sets.
  Arms: Thoracolumbar fascia inhibition group
Other: Suboccipital inhibition group — Soft tissue mobilization: Participants will be asked to lie in a supine position on an appropriate surface and keep their knees in extension. Then, they will be instructed to hold both ends of a sheet and place the middle part of the sheet on the plantar surface of one foot. Using the sheet and by dorsiflexing the ankle, they will pull the extended leg toward themselves. This position should be maintained for 30 seconds (8). It is important that the opposite knee does not flex during the exercise. The application will be performed bilaterally.
  Arms: Suboccipital inhibition group
Other: hamstring stretching — Participants performed passive hamstring stretching using a sheet for self-assistance. Participants will be asked to lie supine on an appropriate surface and keep their knees in extension. Then, they will be instructed to hold both ends of a sheet and place the middle part of the sheet on the plantar surface of one foot. Using the sheet and performing ankle dorsiflexion, they will pull the leg-kept in knee extension-toward themselves. This position should be held for 30 seconds (8). It is important that the opposite knee does not move into flexion during the exercise. The application will be performed bilaterally.

SUMMARY:
This randomized controlled trial aimed to compare the immediate effects of two self-myofascial release techniques-suboccipital muscle inhibition and thoracolumbal fascia inhibition-on hamstring flexibility, spinal range of motion, and balance in healthy adults. A total of 75 participants with hamstring tightness were randomly assigned to one of three groups: suboccipital inhibition, thoracolumbal inhibition, or control. All participants performed hamstring stretching, and the intervention groups received one of the inhibition techniques immediately after. Outcomes were measured at baseline and within 30 minutes post-intervention. The study found that both techniques led to significant improvements in hamstring flexibility and spinal mobility, with region-specific benefits. The thoracolumbal technique was more effective for trunk and hamstring flexibility, while the suboccipital technique provided greater cervical mobility gains. Balance improvements were limited. These findings support the use of targeted myofascial interventions in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between the ages of 18 and 25
* Hamstring muscle tightness as defined by Active Knee Extension Test (AKET) ≥ 20°
* Ability to follow study instructions and provide informed consent
* No participation in other clinical studies within the last 3 months

Exclusion Criteria:

* AKET < 20° (i.e., no hamstring tightness)
* History of musculoskeletal, neurological, or systemic diseases affecting balance or flexibility
* Recent injury or surgery involving the spine, pelvis, or lower extremities
* Use of medications affecting muscle tone or balance
* Inability to perform the required movements or assessments
* Pregnancy or suspected pregnancy

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2025-03-28 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
Change in Cervical Range of Motion (degrees) from Baseline to Post-Intervention | Baseline and immediately (within 30 minutes) post-intervention
  Cervical range of motion (flexion, extension, lateral flexion, rotation) in healthy individuals with hamstring tightness.
Change in Finger-to-Floor Distance from Baseline to Post-Intervention | Baseline and immediately (within 30 minutes) post-intervention
  Finger-to-Floor Distance was used to assess hamstring flexibility. Measurements were taken pre-intervention and within 30 minutes following the intervention.
Change in Y Balance Test from Baseline to Post-Intervention | Baseline and immediately (within 30 minutes) post-intervention
  The Y Balance Test was used to assess dynamic balance, with participants reaching in the anterior, posteromedial, and posterolateral directions while standing on one leg. The average reach distance in centimeters (cm) was recorded for each direction.
  The test was administered at baseline and within 30 minutes post-intervention to assess immediate changes in balance performance.
Change in Active Knee Extension Angle (degrees) from Baseline to Post-Intervention | Baseline and immediately (within 30 minutes) post-intervention
  Active Knee Extension Test (AKET): Degree of knee extension measured using a goniometer. Higher values indicate greater flexibility.
Change in The Stork Balance Test from Baseline to Post-Intervention | Baseline and immediately (within 30 minutes) post-intervention
  The Stork Balance Test was used to evaluate static balance by measuring how long (in seconds) a participant could maintain a balanced stance on one leg.
Change in Lumbal Range of Motion (degrees) from Baseline to Post-Intervention | Baseline and immediately (within 30 minutes) post-intervention
  Lumbal range of motion (flexion, extension) in healthy individuals with hamstring tightness.

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit Üniversity, Kozlu, Zonguldak Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All procedures involving human participants were conducted in accordance with ethical standards. Written informed consent was obtained from all participants prior to the study. Data other than the participants' personal information (e.g., pre- and post-intervention muscle flexibility measurements) were used solely for research purposes. Participant privacy and confidentiality were strictly protected throughout the study.
Supporting Information: Study Protocol, SAP